CLINICAL TRIAL: NCT06092593
Title: Evaluation of Upper Gastrointestinal Tract Lesions in Ulcerative Colitis Patients in Assiut University
Brief Title: Upper Endoscopy in Ulcerative Colitis Patients in Assiut University
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gamal Abdelnasser Gaber Ahmed, Principal investigator, Assiut University
Other Study IDs: Upper endoscopy UC
Record Dates: First submitted 2023-09-28; First posted 2023-10-23 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Upper Gastrointestinal Disorder
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Upper endoscopy — Evaluation of upper gastrointestinal tract lesions in ulcerative colitis patients

SUMMARY:
Aim of study:

Primary Outcomes:

Patients with ulcerative colitis-associated upper gas- trointestinal inflammation may require specific treat- ment for the gastroduodenal lesions. Hence, recogni- tion and detection of the upper gastrointestinal lesions are important. Here we describe 2 cases of ulcerative colitis and summarize the results of our investigation of the prevalence of upper gastrointestinal involvement detected by esophagogastroduodenoscopy. We also analyzed the macroscopic and microscopic features of the upper gastrointestinal lesions

Secondary Outcomes:

correct and timely treatment of upprt GIT lesions in UC .

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is an idiopathic, chronic, relapsing inflammatory bowel disease (IBD) occurring in the colon and rectum . The main typical symptoms of UC include frequent bowel movement, mucus pus, bloody diarrhea, abdominal pain and discomfort, urgency, weight loss, and tenesmus . Apart from these typical symptoms, emerging evidence supports that there are a variety of accompanying symptoms involving the upper gastrointestinal (UGI) tract in patients with UC upon macroscopic and microscopic analyses, such as eosinophilic esophagitis[9], gastroduodenitis, ulcers, or UGI inflammation In addition, the positive rate of UGI endoscopy in asymptomatic individuals was lower than that in symptomatic patients. The reported clinically significant UGI lesions include multiple erosions, granular changes, white spots, friable mucosa, ulcer, and purulent deposits during fibrogastroduodenoscopy (FGDS)[ط UGI involvement may be unnoticed by the attending physician due to the lack of the knowledge of gastroduodenal lesions, which should raise concerns during UC treatment. Furthermore, there is no established standard or criteria available for patients with UC who should undergo FGDS , because the clinical backgrounds of these patients with UC-associated UGI lesions have not been fully and exactly demonstrated. Specific management may be required for patients with UC-associated UGI lesions. Henceforth, we conducted this study with the aim of describing various UGI tract presentations in UC and their differential diagnosis

ELIGIBILITY:
Inclusion Criteria:

* Patients' age is 18 years or above.
* Patient who are diagnosed with UC..
* Patient who are fit to undergo upper endoscopy .

Exclusion Criteria:

* Pediatric patients.
* patient refuse to participate at this study
* patient with known upper GIT disorder .

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A cross sectionaql study will be conducted in Assuit University hospital .Adult patients diagnosed as UC by clinical date , laboratory ,colonscopy and histopathological examination will undergo :
  full medical history taking : age, gender, time since the ulcerative colitis diagnosis, History of surgery for ulcerative colitis, medications , history of any upper GIT symptoms nausea , vomiting , epigastric pain , heart burn , dysphagia and hematemsis or melena .
  complete physical examination , with focus on pulse, blood pressure, body temperature and signs of extra intestinal involvement.
  Esophagogastro-duodenoscopy Histopathological examination of biopsies taken from any lesions
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of upper gastrointestinal tract lesions in ulcerative colitis patients | Baseline
  The relationship between ulcerative colitis patients and upper gastrointestinal tract lesions

REFERENCES:
- [Background] Sun Y, Zhang Z, Zheng CQ, Sang LX. Mucosal lesions of the upper gastrointestinal tract in patients with ulcerative colitis: A review. World J Gastroenterol. 2021 Jun 14;27(22):2963-2978. doi: 10.3748/wjg.v27.i22.2963. PMID 34168401
- [Background] Kato R, Iwamuro M, Hiraoka S, Takashima S, Inokuchi T, Takahara M, Kondo Y, Tanaka T, Okada H. Evaluation of the Upper Gastrointestinal Tract in Ulcerative Colitis Patients. Acta Med Okayama. 2018 Apr;72(2):105-113. doi: 10.18926/AMO/55850. PMID 29674758
- [Background] Queliza K, Ihekweazu FD, Schady D, Jensen C, Kellermayer R. Granulomatous Upper Gastrointestinal Inflammation in Pediatric Ulcerative Colitis. J Pediatr Gastroenterol Nutr. 2018 Apr;66(4):620-623. doi: 10.1097/MPG.0000000000001771. PMID 28991840